CLINICAL TRIAL: NCT05388916
Title: A Real-world, Prospective, Multicenter Study to Assess the Safety and Effectiveness of Secukinumab (Cosentyx®) in Patients Aged 6 to Less Than 18 Years With Moderate to Severe Chronic Plaque Psoriasis in China
Brief Title: A Real-world Study to Assess Safety and Effectiveness of Secukinumab in Pediatric Plaque Psoriasis Patients in China
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457A2406
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Moderate to Severe Chronic Plaque Psoriasis
Keywords: chronic plaque psoriasis; China; NIS; Cosentyx; secukinumab
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cosentyx: Pediatric patients with moderate to severe plaque psoriasis treated with Cosentyx
  Interventions: Other: Cosentyx

INTERVENTIONS:
Other: Cosentyx — Prospective observational cohort study. There was treatment allocation.

SUMMARY:
This was a non-interventional, prospective, multi-center real world setting study, aiming to provide safety and effectiveness data in Chinese pediatric patients with moderate to severe plaque psoriasis treated with Cosentyx® for up to 52 weeks.

DETAILED DESCRIPTION:
Patients who were about to initiate Cosentyx® or had started Cosentyx® within the last 4 weeks and met the eligibility criteria were enrolled. Patients were followed via routine visits in real clinical practice up to 52 weeks. Data from medical records, including safety and effectiveness information of Cosentyx® (e.g., AE, SAE, physical examinations, laboratory tests, disease assessments, etc.) were collected at each visit. No additional study visits, examinations, laboratory tests or procedures were mandated throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting all of the following criteria are eligible for inclusion in this study:

* Written assent and informed consent must be obtained as per local regulations prior to any study procedures.
* Diagnosed with moderate to severe plaque psoriasis.
* Initiating treatment with Cosentyx® or having started Cosentyx® treatment within the last 4 weeks in routine clinical practice, and its prescription is independent of this study.
* Aged 6 to less than 18 years at the time they are prescribed Cosentyx®.
* Have valid PASI and IGA mod 2011 score at the time they are prescribed Cosentyx®.

Exclusion Criteria:

Patients meeting any of the following criteria are not eligible for inclusion in this study:

* Patients previously treated with other biologics.
* Patients participating in other clinical trials or who previously participated in clinical trials within 30 days before Cosentyx® initiation or a period of 5 half-lives of the investigational drug, whichever is longer.
* Patients in conditions which in the judgment of the clinical investigator renders the patient unsuitable for the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Chinese pediatric patients aged between 6 to less than 18 years and diagnosed with moderate to severe plaque psoriasis.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
AEs/SAEs/AESIs type and frequency | 52 weeks
  Adverse events (AEs)/ Serious adverse events (SAEs)/Adverse events of special interest (AESIs).

SECONDARY OUTCOMES:
Percentage of patients who achieved PASI 75 response | Week 12
  Percentage of participants who achieve 75% reduction in the Psoriasis Area and Severity Index (PASI) score compared to baseline. A PASI score is a tool used to measure the severity and extent of psoriasis. The score ranges from 0 (no signs of psoriasis) to a theoretic maximum of 72. The intensity of redness, thickness and scaling of the psoriasis is assessed as none (0), mild (1), moderate (2), severe (3) or very severe (4).
Percentage of patients who achieved IGA mod 2011 0 or 1 response | Week 12
  The Investigator's Global Assessment (IGA) mod 2011 scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and is not compared with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe.
Percentage of patients who achieved PASI 90/100 response | Week 12
  Percentage of participants who achieve 90/100% reduction in the Psoriasis Area and Severity Index (PASI) score compared to baseline. A PASI score is a tool used to measure the severity and extent of psoriasis. The score ranges from 0 (no signs of psoriasis) to a theoretic maximum of 72. The intensity of redness, thickness and scaling of the psoriasis is assessed as none (0), mild (1), moderate (2), severe (3) or very severe (4).
Percentage of patients who achieved PASI 75/90/100 response/IGA mod 2011 0 or 1 response over time | Up to week 52
  Percentage of participants who achieve 75/90/100% reduction in the Psoriasis Area and Severity Index (PASI) score compared to baseline. A PASI score is a tool used to measure the severity and extent of psoriasis.
  The Investigator's Global Assessment (IGA) mod 2011 scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and is not compared with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe.
Absolute value change from baseline of PASI score over time | Up to week 52
  Psoriasis Area and Severity Index (PASI) score s a tool used to measure the severity and extent of psoriasis. The score ranges from 0 (no signs of psoriasis) to a theoretic maximum of 72. The intensity of redness, thickness and scaling of the psoriasis is assessed as none (0), mild (1), moderate (2), severe (3) or very severe (4).
Absolute value change from baseline of IGA mod 2011 score over time | Up to week 52
  The Investigator's Global Assessment (IGA) mod 2011 scale scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- China (7):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18397